CLINICAL TRIAL: NCT06640426
Title: Messaging Intervention to Increase Medicare Annual Wellness Visits: The MIMA Randomized Clinical Trial
Brief Title: Messaging Intervention to Increase Medicare Annual Wellness Visits -- The NUDGE AWV Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emily Rosenzweig (Industry)
Responsible Party: Sponsor-Investigator, Emily Rosenzweig, Director of Behavioral Science, Ascension Health
Organization: Ascension Health (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: RAS20240013
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Annual Wellness Visit; Breast Cancer Screening; Colon Cancer Screening

STUDY DESIGN:
Intervention Model Description: This study will use a randomized controlled trial to evaluate a health system initiative to improve Medicare Annual Wellness Visit (AWV) completion. Investigators will randomly assign Ascension Health patients who are eligible for an AWV to one of three conditions. Patients in Treatment Condition #1 will receive a set of up to five email and text messages over the course of eight days, while also receiving usual care which could include messaging from their practice or the electronic health record. Patients in Treatment Condition #2 will receive a set of two email and text messages on a single day. Patients in the Control Condition will receive no messages as part of this campaign, but will be receiving usual care, which could include messages related to AWV's from their primary care practice or from the electronic health record.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Usual Care (No Intervention): This is a group will serve as usual care and have no intervention during the study period
- Two Messages (Experimental): This group will receive two messages as part of the study -- one email and one text message.
  Interventions: Behavioral: Two Messaging Nudges
- Up To Five Messages (Experimental): This group will receive up to five messages as part o the study -- two emails and three text messages.
  Interventions: Behavioral: Five messaging nudges

INTERVENTIONS:
Behavioral: Two Messaging Nudges — This intervention involves receiving one personalized email and one personalized text message, which include the provider's name, the patient's name, and a phone number to schedule an Annual Wellness Visit
  Arms: Two Messages
Behavioral: Five messaging nudges — This intervention involves patients receiving up to five personalized email and text messages, which include the provider's name, the patient's name, and a phone number to schedule an Annual Wellness Visit
  Arms: Up To Five Messages

SUMMARY:
Medicare Annual Wellness Visits (AWVs) are critical for addressing preventive care needs among older adults, yet the most recent estimates from the Center for Medicare Services suggest less than 50% of eligible patients take advantage of this free healthcare benefit. Behavioral science-informed messaging interventions offer a promising strategy to increase AWV participation by guiding patient behavior. In this study, investigators will evaluate a health system initiative that utilizes personalized email and text messages to encourage Medicare beneficiaries to schedule and attend their AWVs. This approach aims to boost patient engagement in preventive health services, ultimately improving care outcomes for older adult populations

DETAILED DESCRIPTION:
The Centers for Medicare & Medicaid Services (CMS) recommends Annual Wellness Visits (AWVs) to encourage preventive care and improve long-term health outcomes for Medicare beneficiaries. These visits are designed to provide a proactive approach to healthcare by focusing on identifying risk factors, updating medical histories, and developing personalized prevention plans that promote early detection of diseases. By prioritizing prevention over treatment, AWVs help reduce the overall cost burden on the healthcare system while enhancing patient engagement and empowering individuals to take a more active role in managing their health. Yet despite these benefits, most Medicare members who are eligible for an AWV - at no cost to them - do not complete one.

Behavioral science research suggests that personalized messages, designed to facilitate action, can have significant impacts on health behavior. Studies have found these messaging interventions can increase vaccination rates, cancer screening rates, and other care gap closure.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or older
* Have either a mobile phone number or an email address on file with the health system
* Included in and non-compliant on the Ascension AWV Clinical Priority Goal measure
* Have consented to receive electronic communications from the health system

Exclusion Criteria:

* Patients whose primary care providers are exempted from the campaign by the health system
* Completed MAWV appointment in previous 30 days
* Has an upcoming AWV appointment scheduled
* Have received a nudge campaign from the Clinical Transformation team in the past 90 days
* Patients who have previously opted out of receiving electronic communications from the health system in our message delivery platform (Salesforce)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 29842 (Actual)
Dates: Start 2024-10-22 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2025-04-27 (Actual)

PRIMARY OUTCOMES:
Annual Wellness Visit scheduling | 14 days
  Percentage of patients who schedule an AWV

SECONDARY OUTCOMES:
Completed Annual Wellness Visit | 90 Days
  Percentage of patients who have completed an AWV
Days to Annual Wellness Visit Completion | 90 days
  Number of days to AWV appointment completion

OTHER OUTCOMES:
Breast cancer screening | 180 days
  Completion of breast cancer screening post intervention
Colon Cancer Screening | 180 days
  Completion colon cancer screening post intervention
Ordering of tests for breast cancer screening | 90 days
  Ordering of tests for breast cancer screening
Ordering of tests for colon cancer screening | 90 days
  Ordering of tests for colon cancer screening

CONTACTS AND LOCATIONS:
Locations (1):
- Ascension Health, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Has patient information that we are not approved to share